CLINICAL TRIAL: NCT05085808
Title: Comparison of Trazodone vs Quetiapine vs Placebo for the Treatment of ICU Delirium: A Randomized Controlled Trial (The TraQ Study)
Brief Title: RCT: Trazodone vs Quetiapine vs Placebo for Treating ICU Delirium (TraQ)
Acronym: TraQ
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Catherine Kuza, MD, Assistant Professor of Anesthesiology and Critical Care, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APP-20-01962
Record Dates: First submitted 2021-09-27; First posted 2021-10-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Delirium; Morality; Quality of Life; Psych; Treatment Side Effects
Keywords: delirium; quetiapine; trazodone; critical care; ICU delirium
MeSH Terms: conditions — Delirium | interventions — Trazodone; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only unmasked participant will be the pharmacist (who is not part of the study) who will be preparing and packaging the 3 different study medications. The intensivist, ICU RN, patients, patient's family members/legal representative, and additional study personnel will be masked to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Quetiapine (Active Comparator): Start study medication at 25 mg daily PO ; may increase to BID or TID if RASS>=2 or rescue medication must be given; thereafter, if med is TID, dose can be increased by increment of 50 mg q12 hr if RASS>=2 and/or >1 dose of rescue medication is given within 24 hours [max dose 200 mg/day]
  * dose can be reduced/discontinued per discretion of ICU attending if delirium improving, patient experiences AE likely related to study drug, after 14 days of treatment, or patient is discharged from ICU
  * dose should be held if RASS is -3 to -5/comatose/unresponsive or sudden acute change in mental status
  Interventions: Drug: Quetiapine
- Trazodone (Experimental): Start study medication at 25 mg daily PO ; may increase to BID or TID if RASS>=2 or rescue medication must be given; thereafter, if med is TID, dose can be increased by increment of 50 mg q12 hr if RASS>=2 and/or >1 dose of rescue medication is given within 24 hours [max dose 200 mg/day]
  * dose can be reduced/discontinued per discretion of ICU attending if delirium improving, patient experiences AE likely related to study drug, after 14 days of treatment, or patient is discharged from ICU
  * dose should be held if RASS is -3 to -5/comatose/unresponsive or sudden acute change in mental status
  Interventions: Drug: Trazodone
- Placebo (Placebo Comparator): Start study medication at 25 mg daily PO ; may increase to BID or TID if RASS>=2 or rescue medication must be given; thereafter, if med is TID, dose can be increased by increment of 50 mg q12 hr if RASS>=2 and/or >1 dose of rescue medication is given within 24 hours [max dose 200 mg/day]
  * dose can be reduced/discontinued per discretion of ICU attending if delirium improving, patient experiences AE likely related to study drug, after 14 days of treatment, or patient is discharged from ICU
  * dose should be held if RASS is -3 to -5/comatose/unresponsive or sudden acute change in mental status
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trazodone — Trazodone will be administered to ICU patients who need pharmacological intervention for delirium, if they are randomized to the trazodone arm.
  Other Names: Desyrel
  Arms: Trazodone
Drug: Quetiapine — Quetiapine will be administered to ICU patients who need pharmacological intervention for delirium, if they are randomized to the quetiapine arm.
  Other Names: Seroquel
  Arms: Quetiapine
Drug: Placebo — Placebo will be administered to ICU patients who need pharmacological intervention for delirium, if they are randomized to the placebo arm.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the effectiveness of trazodone as compared to quetiapine and placebo, in the management of ICU delirium in adult (>=18 years old) surgical ICU patients. The investigators will compare outcomes such as delirium incidence and duration, in-hospital mortality, 28-day mortality, hospital length of stay (LOS), ICU LOS, mechanical ventilator days, complications, adverse effects, rescue medication use, delirium symptom severity, sleep duration, and sleep quality among participants receiving trazodone, quetiapine, or placebo. The investigators hypothesize participants receiving trazodone will have a shorter duration of delirium, decreased delirium severity, and improved sleep quality compared to participants receiving quetiapine and placebo.

DETAILED DESCRIPTION:
This is a single-center, double-blind randomized, placebo-controlled pilot trial comparing trazodone, quetiapine, and placebo for the treatment of ICU delirium in adult patients admitted to the surgical ICU at Keck Hospital of the University of Southern California.

The purpose of this study is to determine the effectiveness of several medications (trazodone, quetiapine and placebo) used for the treatment of ICU delirium, and their effects on patient outcomes. Since the incidence of ICU delirium is high and has profound negative ramifications on survival, long-term outcomes, cognitive function, in addition to placing a heavy burden on the healthcare system resources and costs, effective delirium treatment strategies are desperately needed. Trazodone is a medication that has promise in delirium treatment, but there is currently insufficient literature to recommend its routine use. The investigators' main objective is to determine if trazodone is an effective and safe treatment option for the management of ICU delirium, and if it results in shorter delirium duration and improved outcomes compared to participants receiving quetiapine and placebo.

Subject screening:

All patients will be screened for study eligibility daily on rounds throughout the study period. Patients eligible for the study will be asked for written informed consent (signed by either the patient or the surrogate decision maker) after admission (even if the patient does not have delirium), or at any point during the ICU course (patient may or may not have a delirium diagnosis at the time of consent).

ICU nurses will assess all patients for delirium at least every 12 hours, using the CAM-ICU tool , in accordance with the standard of care in the surgical ICU (that is, this assessment would be performed regardless of the study).

Patients who have written informed consent, have a diagnosis of delirium (CAM-ICU positive) that requires pharmacological intervention as determined by the attending intensivist, and meet all inclusion criteria and have no exclusion criteria, will be randomized to receive either trazodone, quetiapine, or placebo.

Stratification/Randomization Scheme: Patients who are enrolled in the study, meet randomization inclusion criteria, and have no exclusion criteria, and require a medication intervention for the treatment of ICU delirium, as determined by the attending ICU physician, will be randomized to one of three study arms: 1. Trazodone; 2. Quetiapine or; 3. placebo.

Enrolled patients will be randomized in a 1:1:1 ratio to the Trazodone, Quetiapine, or placebo groups. Randomization will be stratified on age (< vs. ≥65) and delirium severity and occur in blocks, with block size not revealed to investigators. An independent statistician from the USC Clinical and Translational Science Institute (CTSI), will generate a randomization list and import it to REDCap prior to study initiation. Upon confirmation of informed consent, trial eligibility and completion of the baseline assessment, the patient will be randomized to one of the study arms using the REDCap randomization module.

Upon randomization, an automated email notification will be sent to the un-blinded pharmacist (who is not part of the study team), who securely accesses the randomization module on REDCap and will prepare numbered supplement bottles according to the randomization list. The pharmacist will assign and dispense the drug to the ICU nurse who is administering the drug (and is blinded to the medication). The rest of the study team (PIs, co-PIs, research assistants, ICU nurses) will be blinded to the therapy being received and they will be blinded to the randomization and allocation process on REDCap as well, as the allocation and randomization files will be blinded and securely kept under passcode protection by the independent pharmacist. The patients will not know which study medication they are receiving. USC Plaza Pharmacy will prepare the study medications and packaging prior to study initiation.

Study Medication Administration:

There will be standardized method delineating how to begin dosing the study medication, and how to adjust the dose and frequency as needed. Additionally, there will be standardized tapering protocol, so there is consistency among all participants. Furthermore, there will be a standardized rescue medication protocol in place, should patients who are receiving placebo, or having break through delirium despite intervention.

Statistics/Analysis Plan:

-Determination of sample size: As this is a pilot study, a total sample size of 30 (10 per treatment group) over an enrollment period of 1 year is estimated to be recruited based on feasibility. As the primary goal of this pilot study is to identify a signal for treatment efficacy, sample size considerations are based on the precision (i.e., 95% confidence interval) with which key trial parameters can be estimated.

-Baseline descriptive statistics: Baseline characteristics of the study population will be presented by treatment group using conventional descriptive statistics methods, including proportions for categorical variables and means and standard deviations or medians and interquartile ranges for continuous variables, as appropriate based on the data distribution. Comparisons of baseline variables will be performed between treatment groups by one-way Analysis of Variance (ANOVA) for continuous variables and chi-square or Fisher's exact tests for categorical variables, as appropriate. If a statistically significant difference is found (p<0.05) in the ANOVA models, pairwise treatment comparisons will be performed using Tukey's multiple comparison adjustment. Assumptions of the ANOVA model will be tested including 1) normality of model residuals, 2) homogeneity of variance, and 3) independence of observations and if not met, the non-parametric equivalent Kruskal-Wallis test will be used.

-Analysis of primary endpoints: The primary outcome is the duration of ICU delirium measured in days. Differences in the duration of delirium between treatment groups will be analyzed by Poisson regression or negative binomial regression if there is evidence of over-dispersion. Patients with delirium episodes lasting less than one day will be classified as zero days. All models will include the randomized group and randomization stratification variables as independent variables. Model coefficients for each treatment group will be exponentiated to give the estimated rate ratio of each treatment comparison, with 95% confidence intervals. The referent group for treatment group comparisons will be the placebo group (i.e., comparing trazodone to placebo, and quetiapine to placebo). The pairwise comparison of trazodone to quetiapine will also be conducted.

-Analysis of secondary endpoints: Binary secondary endpoints include the proportion of patients with in-hospital mortality, 28-day mortality, who experience complications, and who use rescue medications. The proportion in each treatment group will be compared univariately by the chi-square or Fisher's exact test and in a multivariable model by binary logistic regression.

Additional secondary endpoints include the length of hospital stay, length of ICU stay, and duration of mechanical ventilation (if applicable). These outcomes will be analyzed as described in the "analysis of primary endpoint".

Trial outcomes that are measured daily (delirium severity measured by CAM-S, nightly sleep duration (hours), number of times awoken at night, and sleep quality (Richards Campbell Sleep Questionnaire) will be compared among treatment groups using generalized linear mixed effects models (GLMMs). Normally distributed continuous outcomes will use a normal random outcome with an identify link function; count outcomes (e.g., number of times awoken) will use a Poisson random variable with a log link function. For each model, the primary independent variables will be randomized treatment group and randomization stratification variables. Assessment time (day of assessment, from day 0 to 14) will be treated as indicator variables. The main effect of treatment will estimate the mean of the outcome among treatment groups over the treatment period. An interaction term of treatment-by-day will be used to estimate treatment group means (with SEs and confidence intervals) by intervention day.

-Analysis of safety measures: Numbers and percentages of adverse events and serious adverse events will be cross-tabulated and summarized descriptively by treatment group. No formal statistical analysis will be conducted.

-Populations for analysis: The full analysis dataset will be based on an intention-to-treat (ITT) principle and will be comprised of all study participants who have been randomized to any of the 3 treatment groups. Analysis will be based on the original intervention, regardless of actual intervention received.

ELIGIBILITY:
Inclusion Criteria:

1. >=18-years-old
2. Admitted to the surgical ICU for >24 hours
3. Written informed consent obtained from the patient or their surrogate decision maker.
4. Diagnosis of ICU delirium defined by positive CAM-ICU score AND exhibiting symptomatic delirium (i.e., combative, pulling at lines, a danger to self or others, inability to sleep, hallucinations, etc.), thus, requiring the need for pharmacologic intervention as determined by the attending intensivist

Exclusion Criteria:

1. Acute alcohol or substance abuse withdrawal symptoms/syndrome (i.e., delirium tremens) requiring treatment/intervention (i.e., implementation of the Clinical Institute Withdrawal Assessment for Alcohol (CIWA) protocol, benzodiazepines, alpha-2 agonist, etc.)
2. Recent torsade de pointes or ventricular arrhythmia
3. Prolonged QTc syndrome AND/OR prolonged QT-interval (QTc>500 ms on baseline EKG, performed on the day of randomization)
4. Active psychosis
5. Patients taking medications with known interactions with either trazodone and/or quetiapine
6. Acute encephalopathy (i.e., hepatic, uremic, etc.)
7. Seizure disorder
8. myocardial infarction (MI) within the past 30 days
9. Tardive dyskinesia
10. Hyponatremia
11. Terminal state
12. Diagnosis of liver disease
13. Patients who are strict NPO, are a high aspiration risk (defined as frequent nausea/vomiting, ileus, gastric dysmotility disorder, uncontrolled GERD, weakness/deconditioning, diabetes with gastroparesis, not tolerating full tube feeds if being enterally fed (high residual gastric volume >500 cc), elderly patients with waxing/waning mental status), have dysphagia, and/or have difficulty swallowing capsules as determined by speech therapist
14. Patients who have enteral access such as a small-bore feeding tube, nasogastric or orogastric tube, or gastrostomy/gastrojejunostomy tube (as these patients will need medications crushed in order to administer via the tube, and the capsules used in this study cannot be crushed)
15. Presence of an acute neurologic condition (i.e., acute cerebrovascular accident, intracranial tumor, traumatic brain injury, etc.) on ICU admission. History of stroke or other neurological condition(s) without cognitive impairment is not an exclusion criterion.
16. Pregnancy/lactation
17. History of ventricular arrhythmia including torsade de pointes
18. Allergy/hypersensitivity reaction to trazodone and/or quetiapine
19. Diagnosis of dementia
20. History of neuroleptic malignant syndrome and/or serotonin syndrome
21. Diagnosis of Parkinson's disease or parkinsonism (also referred to as hypokinetic rigidity syndrome)
22. Schizophrenia or other psychotic disorder
23. Patients in whom CAM-ICU cannot be performed to screen for delirium (i.e., acute encephalopathy, mental retardation, vegetative state/coma, deaf, blind, etc.)
24. Inability to speak or understand English
25. Expected to die or transfer out of the ICU within 24 hours
26. Currently enrolled and participating in another interventional study
27. No signed written informed consent by patient or their surrogate decision maker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Delirium duration using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) tool | 14 days
  days

SECONDARY OUTCOMES:
ICU length of stay | 14 days
  days
hospital length of stay | 14 days
  days
mechanical ventilator duration | 14 days
  days
in-hospital mortality | 14 days
  yes or no
28-day mortality | 28 days
  yes or no
complications | 14 days
  yes or no
adverse study drug-related reactions | 14 days
  yes or no
Use of rescue medications | 14 days
  yes or no
Delirium severity | 14 days
  0-19 points using the CAM-S long form
sleep quality | 14 days
  using Richards Campbell Sleep Questionnaire
discharge disposition | 14 days
  home, acute facility, rehabilitation, death, etc.
Long-term cognitive function | up to 6 months post-randomization (measured at 1-, 3-, 6-months post-randomization)
  using MoCA questionnaire
Long-term depression | up to 6 months post-randomization (measured at 1-, 3-, 6-months post-randomization)
  using HADS
Long-term anixety | up to 6 months post-randomization (measured at 1-, 3-, 6-months post-randomization)
  using HADS
Long-term PTSD | up to 6 months post-randomization (measured at 1-, 3-, 6-months post-randomization)
  using IES-R
Long-term quality of life | up to 6 months post-randomization (measured at 1-, 3-, 6-months post-randomization)
  using SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Kuza, MD, FASA, Principal Investigator — University of Southern California
Locations (1):
- Keck Hospital of the University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Kamdar BB, King LM, Collop NA, Sakamuri S, Colantuoni E, Neufeld KJ, Bienvenu OJ, Rowden AM, Touradji P, Brower RG, Needham DM. The effect of a quality improvement intervention on perceived sleep quality and cognition in a medical ICU. Crit Care Med. 2013 Mar;41(3):800-9. doi: 10.1097/CCM.0b013e3182746442. PMID 23314584
- [Background] Reznik ME, Slooter AJC. Delirium Management in the ICU. Curr Treat Options Neurol. 2019 Nov 14;21(11):59. doi: 10.1007/s11940-019-0599-5. PMID 31724092
- [Background] Marra A, Ely EW, Pandharipande PP, Patel MB. The ABCDEF Bundle in Critical Care. Crit Care Clin. 2017 Apr;33(2):225-243. doi: 10.1016/j.ccc.2016.12.005. PMID 28284292
- [Background] Reade MC, Eastwood GM, Bellomo R, Bailey M, Bersten A, Cheung B, Davies A, Delaney A, Ghosh A, van Haren F, Harley N, Knight D, McGuiness S, Mulder J, O'Donoghue S, Simpson N, Young P; DahLIA Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Effect of Dexmedetomidine Added to Standard Care on Ventilator-Free Time in Patients With Agitated Delirium: A Randomized Clinical Trial. JAMA. 2016 Apr 12;315(14):1460-8. doi: 10.1001/jama.2016.2707. PMID 26975647
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Michaud CJ, Bullard HM, Harris SA, Thomas WL. Impact of Quetiapine Treatment on Duration of Hypoactive Delirium in Critically Ill Adults: A Retrospective Analysis. Pharmacotherapy. 2015 Aug;35(8):731-9. doi: 10.1002/phar.1619. Epub 2015 Aug 4. PMID 26238778
- [Background] Mangan KC, McKinzie BP, Deloney LP, Leon SM, Eriksson EA. Evaluating the risk profile of quetiapine in treating delirium in the intensive care adult population: A retrospective review. J Crit Care. 2018 Oct;47:169-172. doi: 10.1016/j.jcrc.2018.07.005. Epub 2018 Jul 5. PMID 30005303
- [Background] Devlin JW, Roberts RJ, Fong JJ, Skrobik Y, Riker RR, Hill NS, Robbins T, Garpestad E. Efficacy and safety of quetiapine in critically ill patients with delirium: a prospective, multicenter, randomized, double-blind, placebo-controlled pilot study. Crit Care Med. 2010 Feb;38(2):419-27. doi: 10.1097/CCM.0b013e3181b9e302. PMID 19915454
- [Background] Devlin JW, Skrobik Y, Riker RR, Hinderleider E, Roberts RJ, Fong JJ, Ruthazer R, Hill NS, Garpestad E. Impact of quetiapine on resolution of individual delirium symptoms in critically ill patients with delirium: a post-hoc analysis of a double-blind, randomized, placebo-controlled study. Crit Care. 2011;15(5):R215. doi: 10.1186/cc10450. Epub 2011 Sep 17. PMID 21923923
- [Background] Knauert MP, Haspel JA, Pisani MA. Sleep Loss and Circadian Rhythm Disruption in the Intensive Care Unit. Clin Chest Med. 2015 Sep;36(3):419-29. doi: 10.1016/j.ccm.2015.05.008. Epub 2015 Jun 29. PMID 26304279
- [Background] Madrid-Navarro CJ, Sanchez-Galvez R, Martinez-Nicolas A, Marina R, Garcia JA, Madrid JA, Rol MA. Disruption of Circadian Rhythms and Delirium, Sleep Impairment and Sepsis in Critically ill Patients. Potential Therapeutic Implications for Increased Light-Dark Contrast and Melatonin Therapy in an ICU Environment. Curr Pharm Des. 2015;21(24):3453-68. doi: 10.2174/1381612821666150706105602. PMID 26144941
- [Background] Pulak LM, Jensen L. Sleep in the Intensive Care Unit: A Review. J Intensive Care Med. 2016 Jan;31(1):14-23. doi: 10.1177/0885066614538749. Epub 2014 Jun 10. PMID 24916753
- [Background] Ishii T et al. Retrospective Study of Trazodone Monotherapy Compared with Ramelteon and Trazodone Combination Therapy for the Management of Delirium. J Psychiatry. 2018; 21(3):1-5
- [Background] Okamoto Y, Matsuoka Y, Sasaki T, Jitsuiki H, Horiguchi J, Yamawaki S. Trazodone in the treatment of delirium. J Clin Psychopharmacol. 1999 Jun;19(3):280-2. doi: 10.1097/00004714-199906000-00018. No abstract available. PMID 10350040
- [Background] Ospina JP et al. Epidemiology, Mechanisms, Diagnosis, and Treatment of Delirium: A Narrative Review. Clinical Medicine and Therapuetics. 2018;1(1):3-9.
- [Background] Popeo DM. Delirium in older adults. Mt Sinai J Med. 2011 Jul-Aug;78(4):571-82. doi: 10.1002/msj.20267. PMID 21748745
- [Background] Wada K, Morita Y, Iwamoto T, Mifune Y, Nojima S. First- and second-line pharmacological treatment for delirium in general hospital setting-Retrospective analysis. Asian J Psychiatr. 2018 Feb;32:50-53. doi: 10.1016/j.ajp.2017.11.028. Epub 2017 Dec 5. PMID 29216606
- [Background] Maeda I, Inoue S, Uemura K, Tanimukai H, Hatano Y, Yokomichi N, Amano K, Tagami K, Yoshiuchi K, Ogawa A, Iwase S; Phase-R Delirium Study Group. Low-Dose Trazodone for Delirium in Patients with Cancer Who Received Specialist Palliative Care: A Multicenter Prospective Study. J Palliat Med. 2021 Jun;24(6):914-918. doi: 10.1089/jpm.2020.0610. Epub 2021 Feb 11. PMID 33577386
- [Background] Berman BD. Neuroleptic malignant syndrome: a review for neurohospitalists. Neurohospitalist. 2011 Jan;1(1):41-7. doi: 10.1177/1941875210386491. PMID 23983836
- [Background] Scotton WJ, Hill LJ, Williams AC, Barnes NM. Serotonin Syndrome: Pathophysiology, Clinical Features, Management, and Potential Future Directions. Int J Tryptophan Res. 2019 Sep 9;12:1178646919873925. doi: 10.1177/1178646919873925. eCollection 2019. PMID 31523132
- [Background] Richards KC, O'Sullivan PS, Phillips RL. Measurement of sleep in critically ill patients. J Nurs Meas. 2000 Fall-Winter;8(2):131-44. PMID 11227580
- [Background] Hodgson C, Needham D, Haines K, Bailey M, Ward A, Harrold M, Young P, Zanni J, Buhr H, Higgins A, Presneill J, Berney S. Feasibility and inter-rater reliability of the ICU Mobility Scale. Heart Lung. 2014 Jan-Feb;43(1):19-24. doi: 10.1016/j.hrtlng.2013.11.003. Epub 2013 Nov 19. PMID 24373338
- [Background] Jones C, Griffiths RD, Humphris G, Skirrow PM. Memory, delusions, and the development of acute posttraumatic stress disorder-related symptoms after intensive care. Crit Care Med. 2001 Mar;29(3):573-80. doi: 10.1097/00003246-200103000-00019. PMID 11373423
- [Result] Jackson P, Khan A. Delirium in critically ill patients. Crit Care Clin. 2015 Jul;31(3):589-603. doi: 10.1016/j.ccc.2015.03.011. Epub 2015 May 4. PMID 26118922
- [Result] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Result] Brummel NE, Girard TD. Preventing delirium in the intensive care unit. Crit Care Clin. 2013 Jan;29(1):51-65. doi: 10.1016/j.ccc.2012.10.007. PMID 23182527
- [Result] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Result] Salluh JI, Latronico N. Making advances in delirium research: coupling delirium outcomes research and data sharing. Intensive Care Med. 2015 Jul;41(7):1327-9. doi: 10.1007/s00134-015-3864-4. Epub 2015 Jun 3. No abstract available. PMID 26077062
- [Result] Zhang H, Lu Y, Liu M, Zou Z, Wang L, Xu FY, Shi XY. Strategies for prevention of postoperative delirium: a systematic review and meta-analysis of randomized trials. Crit Care. 2013 Mar 18;17(2):R47. doi: 10.1186/cc12566. PMID 23506796
- [Result] Ringdal GI, Ringdal K, Juliebo V, Wyller TB, Hjermstad MJ, Loge JH. Using the Mini-Mental State Examination to screen for delirium in elderly patients with hip fracture. Dement Geriatr Cogn Disord. 2011;32(6):394-400. doi: 10.1159/000335743. Epub 2012 Feb 1. PMID 22301509
- [Result] Roberts DJ, Goralski KB, Renton KW, Julien LC, Webber AM, Sleno L, Volmer DA, Hall RI. Effect of acute inflammatory brain injury on accumulation of morphine and morphine 3- and 6-glucuronide in the human brain. Crit Care Med. 2009 Oct;37(10):2767-74. doi: 10.1097/CCM.0b013e3181b755d5. PMID 19865006
- [Result] Collinsworth AW, Priest EL, Campbell CR, Vasilevskis EE, Masica AL. A Review of Multifaceted Care Approaches for the Prevention and Mitigation of Delirium in Intensive Care Units. J Intensive Care Med. 2016 Feb;31(2):127-41. doi: 10.1177/0885066614553925. Epub 2014 Oct 27. PMID 25348864
- [Result] van den Boogaard M, Schoonhoven L, Evers AW, van der Hoeven JG, van Achterberg T, Pickkers P. Delirium in critically ill patients: impact on long-term health-related quality of life and cognitive functioning. Crit Care Med. 2012 Jan;40(1):112-8. doi: 10.1097/CCM.0b013e31822e9fc9. PMID 21926597
- [Result] Davydow DS. Symptoms of depression and anxiety after delirium. Psychosomatics. 2009 Jul-Aug;50(4):309-16. doi: 10.1176/appi.psy.50.4.309. PMID 19687169
- [Result] Breitbart W, Gibson C, Tremblay A. The delirium experience: delirium recall and delirium-related distress in hospitalized patients with cancer, their spouses/caregivers, and their nurses. Psychosomatics. 2002 May-Jun;43(3):183-94. doi: 10.1176/appi.psy.43.3.183. PMID 12075033
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Weiss DS, Marmar CR, Wilson JP, et al. Assessing psychological trauma and PTSD. The Impact of Events Scale. 1997;19:399-411.
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914